CLINICAL TRIAL: NCT02225795
Title: A Pilot Study of Autologous Hematopoietic Stem Cell Transplantation With Post-transplant Cyclophosphamide for Children and Young Adults With Refractory Crohn's Disease.
Brief Title: Pilot Study of Stem Cell Transplantation for Children and Young Adults With Refractory Crohn's Disease.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: TriStar Health (Other)
Responsible Party: Principal Investigator, Haydar Frangoul, Medical Director, Pediatric Hematology Oncology, TriStar Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT 12
Record Dates: First submitted 2014-07-28; First posted 2014-08-26 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Hematopoietic stem cell transplantation; Children; Young Adults
MeSH Terms: conditions — Crohn Disease | interventions — Hematopoietic Stem Cell Transplantation; Antilymphocyte Serum; Cyclophosphamide; Hematopoietic Stem Cell Mobilization; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm: All subjects (Experimental): Hematopoietic stem cell transplantation
  Interventions: Other: Hematopoietic stem cell transplantation

INTERVENTIONS:
Other: Hematopoietic stem cell transplantation — Immuno-ablative regimen for HSCT:
  Day Treatment
  * 6 r-ATG 2 mg/kg
  * 5 r-ATG3 2 mg/kg
  * 4 r-ATG3 2 mg/kg
  * 3 Cyclophosphamide with Mesna
  * 2 Cyclophosphamide with Mesna
  * 1 REST 0 PBSC infusion
    * 3 Cyclophosphamide with Mesna
    * 4 Cyclophosphamide with Mesna
    * 6 Start GCSF
  Other Names: ANTI-THYMOCYTE GLOBULIN (Rabbit) NSC# 720095; CYCLOPHOSPHAMIDE (Cytoxan) NSC #26271; MESNA - INJECTION NSC #113891; GCSF: Filgrastim: 5 mcg/kg iv; Stem-cell mobilization; Leukapheresis

SUMMARY:
This is a study for people with Crohn's Disease (CD) that are not responsive to standard treatment. CD is a chronic disease with an auto-immune component that goes away and relapses over the years and causes lifelong impairment of health and quality of life. Regardless of the therapy used some patients remain seriously ill with active disease after multiple therapeutic options have been exhausted. There is currently no drug that will cure CD. Drug treatment is focused on controlling symptoms. Another treatment is to perform surgery but again this does not lead to cure and is often linked to infection, short gut syndrome problems and psycho-social and cosmetic issues. Therefore, a treatment that does not involve surgery or long-term drug treatment may be beneficial especially to young adults.

Hematopoietic stem cell transplantation (HSCT) has been of value in other auto-immune diseases and it is possible that it could be of value in CD. This is a pilot study to determine if HSCT is safe and effective for children and young adults with severe CD. For this study the stem cells will come from the patient. This is called an autologous transplant. The patient will undergo collection and storage of his/her peripheral blood stem cells (PBSC). The patient will be given drugs to move (or mobilize) the stem cells from his/her bone marrow into his/her blood where they will be collected on a machine called apheresis (similar to dialysis.) The cells will be stored and given back to the patient about 1 month after collection.

DETAILED DESCRIPTION:
Crohn's Disease (CD) is an immunologically mediated chronic illness that has a relapsing and remitting course, most commonly presenting in the 2nd or 3rd decade and causing lifelong impairment of health and quality of life. Mainstay of clinical treatment for severe disease is combination of anti-inflammatory agents like 5-aminosalicyaltes and immunosuppressive medications like corticosteroids and newer anti-TNF antibodies like Infliximab. None of the drugs are, at present, curative and a relevant subset of patients are refractory to many of these pharmacologic approaches.

Immunoablative treatment followed by autologous stem cell rescue (Autologous HSCT) has been tried in this refractory group of patients with successful results. Autologous HSCT is effective in this auto-immune setting through the eradication of effector/memory T-cell clones due to a direct immuno-ablative effect of drugs used in the preparative regimen; by leading to an immune-reset- recovering clones of T- cells from the infused stem cells do not mount an auto- immune response and are tolerant to 'self' antigens and, by upregulation of T regulatory cells (Treg, CD4+CD25+FOXP3+ or CD8+ FOXP3+) via change in cytokine mileu during transplant. Increased population of Tregs restricts the activity of self-reactive effector T-cells.

This pilot study is designed to gain on the success of previously published adult studies of autologous HSCT in refractory CD, with the aim to confirm the feasibility, safety and efficacy of HSCT and post-transplant cyclophosphamide when given post-HSCT in pediatric patients and young adults.

Since, this combination of immuno-ablative therapy with post-transplant cyclophosphamide has not been extensively studied in children with CD, therefore transplant related mortality (TRM) and severe toxicity (> grade 3 toxicity by NCI criteria) will be monitored for 100 days post-transplant in all the patients and stopping rules will be enforced in case of excessive toxicity or TRM (>10%). Clinical assessments will be done for 1 year post-HSCT for disease activity, steroid free remission period to evaluate the 'clinical efficacy' of this procedure.

The major aim of this pilot is to generate the preliminary safety data to confirm the feasibility and benefit of autologous HSCT in children and young adults with refractory CD.

Study Design:

This is a single arm, pilot study designed to estimate the feasibility, safety and benefit of immunoablation with hematopoietic stem cell transplantation (HSCT) using autologous stem cells followed by administration of post-transplant cyclophosphamide for children and young adults with refractory Crohn's disease (CD). The study population is patients with severe and refractory Crohn's disease who are ≥10 and ≤ 30 years of age.

Objectives:

Primary Objective:

To determine the feasibility and toxicity of immunoablation with HSCT and post-HSCT infusion of cyclophosphamide in children and young adults with refractory Crohn's disease (CD). Death (transplant related mortality, TRM) and severe non-hematologic toxicity (≥ grade 3 toxicity; NCI Toxicity Criteria version 4.0) within the first 100 days after HSCT will be monitored to meet this end-point.

Secondary Objectives:

Secondary objectives are evaluations of incidence of HSCT related complications and evaluations of response. These include:

1. Incidence of viral reactivations - CMV and EBV
2. Incidence of invasive fungal infections
3. Immune reconstitution after HSCT lymphocyte subpopulations (absolute number of CD3, CD4, CD8 and CD19 cells), immunoglobulin levels (IgG) and CD4+ CD25+ CD127+ regulatory T cells (Treg) populations on day +30 , +60 , +100, day +180 and yearly post-HSCT.
4. Evaluate the efficacy and benefit of HSCT in this population at 1 year post HSCT, by serial assessments of clinical activity of CD, assessment of disease severity- CDAI scores and length of steroid free remissions.

Hypotheses:

Primary: The HSCT and post-transplant cyclophosphamide regimen will be well tolerated with acceptable toxicity and will lead to <10% transplant related mortality (TRM).

Background and Rationale:

Crohn's disease (CD) is a chronic illness that is immunologically mediated, of unknown etiology, but probably induced by an exposure to intestinal bacteria or their component antigens leading to an excessive T helper type 1 (TH-1) mediated chronic inflammation of the gastrointestinal (GI) tract 1. Crohn's disease is a relapsing and remitting disorder most commonly presenting in the 2nd or 3rd decade and causing lifelong impairment of health and quality of life 2.

Regardless of the therapy used some patients remain seriously ill with active disease after multiple therapeutic options have been exhausted. In addition, patients with refractory disease suffer from an inability to eat, frequent nausea, vomiting, diarrhea, malnutrition, growth retardation, fistulae formation, abdominal pain and psychological distress, ileostomy or colostomy, and multiple surgeries that may lead to short-gut syndrome, severely affecting quality of life. Though not well characterized, a distinct excessive mortality exists in this group of patients 3,4.

Patients with refractory CD have a higher mortality rate compared to normal population (hazard ratio of 1.73); but deaths are usually related to surgical complications, liver disease, infections and intestinal cancer in long term survivors 5. Even though the overall mortality is low in this group of patients, they suffer from significant morbidity, cortico-steroid side effects and poor quality of life and 50% patients with refractory disease will need surgical interventions (ileostomy, colostomy) further affecting the complications rate 2,3.

Many drugs have been used for controlling the symptoms of CD, but no drug is, at present, curative and a relevant subset of patients are refractory to many pharmacologic approaches 6. Almost all drugs employed in the advanced form of disease, such as immunosuppressives and immunomodulators, have potential risks. Mainstay of clinical treatment is combination of anti- inflammatory agents like 5-aminosalicyaltes and immunosuppressive medications like corticosteroids4. Majority of the patients with severe refractory disease are treated with anti- Tumor Necrosis Factor (TNF) antibodies like Infliximab (Remicade), but limited options exist for patients who have failed to respond to anti-TNF therapy7. Approximately 40% of patients with CD develop intolerable side effects or fail to respond to anti-TNF therapy, hence there is a significant population of this subset of patients where options are very limited 8.

Some symptoms may be controlled by prolonged steroids, but there are many known long term effects of continued steroid use- muscle loss, osteopenia, cataracts and cushingoid habitus. Majority of these patients enroll on other experimental Phase I/II drug trials or resort to surgical intervention to control symptoms. Surgical approach (partial gut resection of the inflamed segment with ileo-colostomy) is an option, but is associated with infection risk, psycho-social and cosmetic issues and increased morbidity due to short gut syndrome, especially in young adults. Increased mortality is also associated with surgical interventions 2,3.

Therefore, any intervention that avoids surgery or long term corticosteroids in young adults may be beneficial. Given that hematopoietic stem cell transplantation (HSCT) have been of some value in other auto-immune diseases characterized by loss of immune tolerance and or a TH-1 predominant immune response, it is possible that these procedures could be of value in CD 9,10. Autologous transplantation might also be of benefit because clearing the body of committed lymphocyte clones might restore the patient to the status quo ante of being predisposed to CD but not suffering from it 11.

Rationale of HSCT for CD

HSCT may provide benefit in auto-immune disease by:

1. Eradication of effector/memory T-cell clones due to a direct immuno-ablative effect of drugs used in the preparative regimen.
2. Immune-reset: recovering clones of T-cells from infused stem cells do not mount an auto-immune response and are tolerant to 'self' antigens.
3. Upregulation of T regulatory cells (Treg, CD4+CD25+FOXP3+ or CD8+ FOXP3+) - by change in cytokine mileu during transplant. Increased population of Tregs restricts the activity of self-reactive effector T-cells.
4. Engraftment of uncommitted stem cells in the gut mucosa may lead to direct healing of mucosa.

Evidence for the effectiveness of HSCT in Crohn's disease Initial observations were made in patients with Crohn's disease and hematologic malignancies. For patients who underwent HSCT for their hematologic malignancy they had remission of their Crohn's disease 12.

Several studies have reported the clinical course of patients with Crohn's disease receiving autologous transplantation for another condition. Perhaps the most interesting concerned a patient who developed symptoms at the age of 9, who was diagnosed with Crohn's disease 4 years later and who required substantial treatment over the next 7 years 13. Following autologous stem cell transplantation for non-Hodgkin's lymphoma it was reported that there was no clinical or laboratory evidence of recurrence of his Crohn's disease in the next 7 years. Another reported case of Crohn's disease had diffuse pan colitis before transplantation and was asymptomatic (but had inflammation) at endoscopy 3 years later 14. Another patient who had symptomatic Crohn's disease for 2 years and had undergone surgery was free of disease 5 years after transplantation. Systematic colonoscopic evaluation showed persisting subclinical inflammation initially with progressive clearance. At Vanderbilt we performed an unrelated donor transplant for a patient with AML and Crohn's disease. He is currently 10 years post-transplant with no symptoms of Crohn's disease.

HSCT specifically for Crohn's disease:

The first report of stem cell transplantation for Crohn's disease concerned 2 patients from the Chicago group 15. In both of the initial cases Crohn's disease activity index was more than 250 (normal range <150, pathological range 220 - 600) despite treatment with infliximab. In both patients, peripheral blood stem cells (PBSC) were mobilized using cyclophosphamide and granulocyte colony stimulating factor (G-CSF), enriched ex-vivo by CD 34+ selection. Cyclophosphamide and antithyomcyte globulin (ATG) were used for immune conditioning prior to transplantation. The first patient was a 22 year old woman with a past history of a right hemicolectomy with severe ileocolic Crohn's disease causing intractable diarrhea with 25 bowel actions per day, fistula and peri-anal sepsis. The second was a 16 year old boy who had been unwell for 6 years requiring tube feeding and receiving methotrexate, 6-mercaptopurine and 5 amino acyclic acid with Crohn's colitis. In both of these cases, following transplantation, diarrhea resolved and the Crohn's disease activity index normalized. In the first patient the haemoglobin rose, whereas in the second it remained at a slightly sub-normal level. Post-transplantation CRP was within normal limits and the albumin remained or became normal. These cases were accompanied by extensive colonoscopic evidence of disease activity. Prior to transplantation both cases had areas of severely active Crohn's disease with cobble stoning, fissuring and deep ulceration. Following transplantation the bowel remained abnormal though changes were much more trivial with superficial erosions only.

Oyama et al reported on autologous HSCT for 12 patients median age of 27 (15-38) with severe refractory Crohn's disease 16. The conditioning regimen consisted of cyclophosphamide (200 mg/kg) and equine ATG (90 mg/kg). Eleven of 12 patients entered a sustained remission defined by a CDAI < 150. After a median follow-up of 18.5 months (range, 7-37 months), only one patient has developed a recurrence of active CD, which occurred 15 months after HSCT.

Hasselbatt et al reported on autologous HSCT 12 patients (ages 24-50) with refractory Crohn's disease using high dose cyclophosphamide (200 mg/kg) without ATG 17. PBSC harvest following mobilization chemotherapy was successful in 11/12 patients and resulted in a clinical and endoscopic improvement in 7/12 patients. Subsequent conditioning and autoPBSCT were performed in nine patients and were relatively well tolerated. Among those, five patients achieved a clinical and endoscopic remission within 6 months after autoPBSCT. However, relapses occurred in 7/9 patients during follow-up, but disease activity could be controlled by low-dose corticosteroids and conventional immunosuppressive therapy.

In 2010 Burt et al reports on autologous HSCT in 24 patients with mean age of 24 years (range 15-52) with anti-TNF refractory Crohn's disease 18. Stem cells were mobilized from the peripheral blood using cyclophosphamide (2.0 g/m2) and G-CSF (10 ug/kg/day), enriched ex vivo by CD34 selection, and reinfused after immune suppressive conditioning with cyclophosphamide (200 mg/kg) and either equine antithymocyte globulin (ATG, 90 mg/kg) or rabbit ATG (6 mg/kg). Eighteen of 24 patients are 5 or more years after transplantation. All patients went into remission with a CDAI less than 150. The percentage of clinical relapse-free survival defined as the percent free of restarting CD medical therapy after transplantation is 91% at 1 year, 63% at 2 years, 57% at 3 years, 39% at 4 years, and 19% at 5 years.

The percentage of patients in remission (CDAI < 150), steroid-free, or medication-free at any posttransplantation evaluation interval more than 5 years after transplantation has remained at or greater than 70%, 80%, and 6% respectively.

Regulatory T cells (Tregs) and Auto-immune disease:

Regulatory T cells (Tregs) are implicated in the suppression of immune responses and in maintenance of tolerance 19,20. The percentage of CD4+CD25+FOXP3+ T cells (T regs) is significantly decreased in patients with auto-immune diseases like SLE and Type 1 diabetes 20. Also, transfer of Treg can prevent auto-immune phenotype that develops after Treg depletion in animal models.

During HSCT for auto-immune diseases, an increase in Treg population correlates with remission induction. Zhang et.al has shown that HSCT leads to a newly generated population of Treg cells that maintain patients in true immunological remission 21.

Burt et.al, also evaluated the role of Treg cells in some of their patients who underwent HSCT for CD. Before HSCT the mean % of Treg cells was significantly low in CD patients (2.62% ± 2.01%), compared to normal volunteers (3.86% ± 1.67%). A robust increase in the % of Treg was observed after HSCT, but this was not sustained over period of time and may have contributed to relapses 18. Hence, there is clinical evidence that a sustained increase in Treg population may maintain remission in patients with auto-immune disorder.

Rationale of the proposed Study:

This pilot study is designed to estimate the feasibility of HSCT and safety of post-HSCT cyclophosphamide infusions for patients with refractory disease who have failed to respond to Infliximab/and or other immunosuppressive agents. This is designed as a small pilot study with built in 'stopping rules' in case of excessive toxicity or death.

Rationale for the immuno-ablative regimen:

Rationale of CY for mobilization: Cyclophosphamide (CY) will be used for mobilization of peripheral stem cells and for immuno-ablation prior to HSCT. CY has been traditionally used for mobilization in all HSCT for refractory CD.

Rationale for post-transplant Cyclophosphamide (CY)- Recently, use of post-transplant CY has been pioneered by John Hopkins and shown to be a very effective GVHD prophylaxis in patients undergoing HSCT for hematologic malignancies, even in the setting of HLA mismatched and haploidentical donors. Post-transplant delivery of CY allows for effective deletion of proliferating allo-reactive T- cells that cause GVHD without adding to the toxicity of the regimens 22. In a recent study by the Hopkins group post-transplant cyclophosphamide was successfully used in patients with sickle cell disease undergoing haploidentical bone marrow transplant with no toxicities.

Some studies have performed CD34+ stem cell selections to get rid of all immune-reactive T- cells clones and use purified CD34+ infusions for regenerating the immune system 18. The problem with this approach is delayed immune-reconstitution post-transplant and a higher incidence of infections.

European trials have used un-manipulated peripheral blood stem cells (PBSCs) as infusions (without any T cell depletion or CD34+ selections) for SCT in auto-immune diseases 23. Since, peripheral stem cells contain the same T cells clones that are immuno-reactive and are infused along with the donor stem cells in non-T cell depleted infusion, this may be one of the reasons for relapse in T cell replete HSCT done till date for CD.

Therefore, to overcome the above-mentioned issues, we propose to use un-manipulated PBSCs, but give two doses of CY pre- and two doses post-stem cell infusion to effectively deplete the immuno-reactive T cell clones present in the autologous infusion and therefore, decrease the incidence of relapse. The total dose of CY remains the same (200 mg/kg), therefore, it will not add to the toxicity of the regimen, but may lead to more effective depletion of the immune- reactive clones, obviating the need for costly in-vitro T cell depletions/CD34+ selections.

Also, CY causes sustained depletion of all T cell subsets, but more profound depletion of CD4+ CD25- subsets, resulting in relative enrichment of CD4+CD25+ cells, which we hope to expand by using post-transplant cyclophosphamide.

Rationale for Rabbit-ATG (Thymoglobulin, Genzyme Corp, Cambridge, MA): will also be used for effective immune-ablation and for in-vivo T cell depletion post- stem cell infusion. Rabbit ATG will be used as this has been shown to promote the expansion of functional Tregs in-vitro 24. Rabbit ATG was use in the largest study by Burt et al 18.

(Please note reference numbers can be found on pages 25-26 of the protocol.)

ELIGIBILITY:
Inclusion Criteria:

All the subjects considered eligible for the study will be screened and reviewed by the Gastroenterology (GI) physicians prior to enrollment (Dedrick Moulton, MD or his designee at Vanderbilt Children's Hospital) 2. Age ≥ 10 and < 30 years 3. Disease status:

1. Confirmed diagnosis of Crohn's Disease: Diagnosis of Crohn's disease that has been established based on typical endoscopic/histologic and/or radiological appearances.
2. Active disease, defined as: Pediatric Crohn's Disease Activity Index (PCDAI) >30 (see Appendix I) or Crohn's Disease Activity Index (CDAI) of >250 (see Appendix II) at any time within 3 months prior to enrollment and any one of the following- i. Endoscopic evidence of active disease confirmed on histology within 3 months prior to enrollment, or ii. Clear evidence of active small bowel Crohn's disease on small bowel imaging within 3 months prior to enrollment.
3. Refractory disease- Moderate to severe disease that has been unresponsive to current or prior therapy with mercaptopurine and/or azathioprine (thiopurines), methotrexate and anti-TNF therapy. Patients should have relapsing disease (i.e. ≥ 1 exacerbation/year) or corticosteroid dependence despite current or prior thiopurines, methotrexate and anti-TNF maintenance therapy or clear demonstration of intolerance or toxicity to these drugs. Patients who fail induction therapy with corticosteroids and anti-TNF therapy, and are therefore not eligible to receive maintenance therapy with thiopurines or methotrexate will also be candidates for enrollment.

   4. Negative stool culture, C. difficile, and negative CMV pcr (in stool or colonic biopsy). Patients with CMV colitis will receive a trial of anti-viral treatment and only responders will be considered eligible for inclusion.

   5. Patients with a prior ileostomy or colostomy may enter the study. For this group of patients', physician's global assessment will be used to assess clinical activity of CD, as Pediatric CDAI and CDAI scoring method may not be representative of disease activity.

   6. Patients with abscesses are eligible to enroll once the abscesses or any other significant infection has resolved.

Exclusion Criteria:

1. Pregnancy or unwillingness to use adequate contraception during the study- if a woman is of childbearing age.
2. HIV infection.
3. Organ function criteria-

   1. Renal: creatinine clearance < 50 ml/min/1.73m2 (measured or estimated).
   2. Cardiac: left ventricular ejection fraction <30% by multigated radionuclide angiography (MUGA) or a shortening fraction of < 25% by cardiac echocardiogram.
   3. Pulmonary Function tests: DLCO < 30% or patient on oxygen.
   4. Hepatic: serum bilirubin > 3 mg%; AST and ALT > 3x ULN for the institutional lab.
4. Uncontrolled Hypertension (using age based criteria) despite at least 2 anti- hypertensive agents.
5. Active Infection or risk thereof-

   1. Current abscess or significant active infection
   2. Perianal infection is not an exclusion criterion, provided there is drainage with or without placement of drain.
   3. Abnormal chest x- ray (CXR) consistent with active infection or neoplasm.
6. Severe diarrhea due to short small bowel; patients believed to have < 700 mm of small bowel and diarrhea attributable to this will be excluded.
7. Patients with toxic megacolon, active bowel obstruction or intestinal perforation.
8. Unable to collect minimum of 3 x106/kg CD34+ cell dose. These patients will be excluded from receiving the preparative regimen.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility and toxicity of immunoablation with HSCT and post-HSCT infusion of cyclophosphamide in children and young adults with refractory Crohn's disease (CD). | first 100 days post HSCT
  This is a composite outcome to determine the feasibility and toxicity of immunoablation with HSCT and post-HSCT infusion of cyclophosphamide in children and young adults with refractory Crohn's disease (CD). Death (transplant related mortality, TRM) and severe non-hematologic toxicity (≥ grade 3 toxicity; NCI Toxicity Criteria version 4.0) within the first 100 days after HSCT will be monitored to meet this end-point.

SECONDARY OUTCOMES:
1. Incidence of viral reactivations - CMV and EBV | First 100 days post HSCT
2. Incidence of invasive fungal infections | within first 100 days post HSCT
3. Immune reconstitution after HSCT | Until the study is closed which is anticipated to be approximately 3 years.
  3. Immune reconstitution after HSCT lymphocyte subpopulations (absolute number of CD3, CD4, CD8 and CD19 cells), immunoglobulin levels (IgG) and CD4+ CD25+ CD127+ regulatory T cells (Treg) populations on day +30 , +60 , +100, day +180 and yearly post-HSCT.
4. Evaluate the efficacy and benefit of HSCT in this population at 1 year post HSCT, by serial assessments of clinical activity of CD, assessment of disease severity- CDAI scores and length of steroid free remissions. | 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Haydar Frangoul, MD, Principal Investigator — TriStar Health